CLINICAL TRIAL: NCT04468477
Title: An Evaluation of the Safety and Clinical Utility of Handheld ECG Technology in Cardiology
Brief Title: EVALECGcardio Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CD20/130832
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients attending cardiac outpatient clinic (Active Comparator)
  Interventions: Device: 6 Lead ECG

INTERVENTIONS:
Device: 6 Lead ECG — Patients will be assessed with the Kardiamobile device.

SUMMARY:
ECGs are routinely performed in cardiology. Recently handheld ECGs have shown promise in screening for heart rhythm disorders. These are quick to perform and do not require the preparation that is needed for 12 lead ECGs. We wanted to test whether a novel handheld ECG recorder, Kardia 6L, which has the potential to record a 6 lead ECG is able to screen for ECG abnormalities, thereby obviating the need for a full 12 lead ECG. This may allow for earlier diagnosis and treatment.

DETAILED DESCRIPTION:
The aim of analysis is to determine if the handheld 6 lead ECG can be used as a simple screener to identify patients who do not need a 12 lead ECG.

ELIGIBILITY:
Inclusion Criteria:

* Anyone attending cardiology outpatients or the ward who has had a recent ECG (within 6 hours)

Exclusion Criteria:

* Patients who do not consent to the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2021-05-21 (Estimated); Study Completion 2021-05-21 (Estimated)

PRIMARY OUTCOMES:
Difference between the 6 lead and the 12 lead Electrocardiogram | 2 minutes
  Sensitivity and specificity of handheld 6Lead compared to 12lead for the measurement of the stages of heart rhythms.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom